CLINICAL TRIAL: NCT04654845
Title: Patient Perception Between Two Emergency Treatments of Symptomatic Irreversible Pulpitis. A Randomized Multicenter Clinical Trial.
Brief Title: Patient Perception Between Two Emergency Treatments of Symptomatic Irreversible Pulpitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, DDS, Aula Dental Avanzada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PULP
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Irreversible Pulpitis
Keywords: Pulpotomy; Pulpectomy
MeSH Terms: interventions — Pulpotomy; Pulpectomy

STUDY DESIGN:
Intervention Model Description: Participants with irreversible pulpitis are randomly assigned to one type of intervention.
Who Masked: Participant
Masking Description: The patient will not be aware of the type of procedure he has been assigned for.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulpotomy (Experimental): Only the tissue in the pulp chamber will be removed.
  Interventions: Procedure: Pulpotomy
- Pulpectomy (Active Comparator): Both the chamber´s and root´s pulp tissue will be removed up to a 25 gauge.
  Interventions: Procedure: Pulpectomy

INTERVENTIONS:
Procedure: Pulpotomy — Access to pulp chamber. Removal of the pulp chamber tissue. Use of Sodium Hypochlorite (5.25% NaCl) during the whole procedure and in the amount considered appropriate by each operator.
  Wait until confirmation of absence of bleeding from the conducts. Placement of polytetrafluroethylene in pulp chamber. Placement of temporary filling. Reduction of the occlusal surface of the tooth until there is no contact with the articulating paper from 200μ.
  Arms: Pulpotomy
Procedure: Pulpectomy — Access to pulp chamber. Removal of the pulp chamber tissue. Use of Sodium Hypochlorite (5.25% NaCl) during the whole procedure and in the amount considered appropriate by each operator.
  Establishment of working length by means of Electronic Apex Locator and a number 8 K file.
  Access to all conducts with a number 10 K file. Rotary instrumentation with one reciprocating system up to working length and up to an apical diameter of 25.
  Placement of polytetrafluroethylene in pulp chamber. No intermediate medication will be filled into the conducts.
  Placement of temporary filling. Reduction of the occlusal surface of the tooth until there is no contact with the articulating paper from 200μ.
  Arms: Pulpectomy

SUMMARY:
To evaluate in a comparative way the perception of the patient who comes with pain due to irreversible pulpitis in a tooth and who receives two types of treatment: complete pulpectomy (or control group) or pulpotomy (or experimental group).

Prospective randomized and multicenter study. It will be carried out in 4 centers of similar socio-professional characteristics, with the same operative protocol. On a significant sample of emergency patients with a concrete clinical manifestation of symptomatic irreversible pulpitis, one type of intervention or another will be performed randomly. The data will be collected by means of a visual numeric scale (NRS).

The null hypothesis is that both interventions provide the same reduction of pain in patients who present symptomatic irreversible pulpitis.

All the patients who come to one of the private centers with irreversible pulpitis and who meet the defined criteria for inclusion and exclusion will be selected.

The type of procedure that will be performed in the control group will be the complete removal of the pulp by means of a defined instrumentation technique, also called Pulpectomy. The procedure to be performed in the experimental group will be the removal of the pulp only at coronal level, also called Pulpotomy. The interventions will be assigned randomly and the "List Randomizer" (random.org) will be used for the randomization.

DETAILED DESCRIPTION:
Clinical procedure will be the same in both groups with regard to the anesthetic technique, and the cavity access and provisional closure of the aperture. The characteristics of both interventions will be described in detail in order to homogenize the procedures. The patient will be conveniently informed before requesting his/her Informed Consent for his/her voluntary participation in the study. Their identification data will be treated in accordance with the provisions of Regulation (EU) 2016/679 of the European Parliament and Council of April 27, 2016, and the Organic Law 3/2018 of 5/12, currently in force, will remain in custody at the Center where they receive treatment and will not be shared by the other centers of the study.

The patient will not be aware of the type of procedure he has been assigned for and will express in a numerical scale according to his perception of the pain on 4 occasions: before starting treatment, at 8-12, 24 and 72 hours after treatment. Likewise, right after receiving the treatment, he will answer some questions related to the degree of comfort during the treatment and about his perception of the time of the intervention.

Data sheets will be collected and treated statistically.

ELIGIBILITY:
Inclusion Criteria:

* Patient in American Society of Anesthesiologists I or II condition.
* Patient who comes to the emergency room with irreversible pulpitis in a single tooth.
* Patients of age >20 years.
* Positive response to the vitality test and bleeding after pulp exposure.

Exclusion Criteria:

* American Society of Anesthesiologists patients>II.
* Pharmacological allergies that contraindicate the intervention.
* Teeth with negative vitality test and no bleeding after pulp exposure.
* Signs of concomitant periodontal infection such as swelling or fistula.
* Teeth with immature roots.
* Patients who are medicated with anxiolytics.
* Abuse of psychotropic drugs or medication that may alter the perception of pain 15 days before the intervention.
* Pregnant or breast-feeding women.
* Interventions with conscious sedation.
* Pathological mental state (dementia, psychosis).
* Lack of collaboration or non-acceptance of the consent of the study.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Patients´ pain perception | Through study completion, an average of 1 year.
  The patient's perception of the degree of post-operative pain following emergency treatment

SECONDARY OUTCOMES:
Procedure time | Through study completion, an average of 1 year.
  The time it takes for each procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Esteve-Pardo, DDS, Principal Investigator — Aula Dental Avanzada
Locations (4):
- Spain (4):
  - Clínica Dental 4, Ferrol, A Coruña
  - Clínica Dental Corbalán, Ceutí, Murcia
  - Centro Dental Navarro Ferri, Cullera, Valencia
  - Clínica Dental esteve, Alicante

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gatewood RS, Himel VT, Dorn SO. Treatment of the endodontic emergency: a decade later. J Endod. 1990 Jun;16(6):284-91. doi: 10.1016/S0099-2399(06)81631-6. PMID 2074427
- [Background] Lee M, Winkler J, Hartwell G, Stewart J, Caine R. Current trends in endodontic practice: emergency treatments and technological armamentarium. J Endod. 2009 Jan;35(1):35-9. doi: 10.1016/j.joen.2008.10.007. PMID 19084121
- [Background] Nyerere JW, Matee MI, Simon EN. Emergency pulpotomy in relieving acute dental pain among Tanzanian patients. BMC Oral Health. 2006 Jan 21;6:1. doi: 10.1186/1472-6831-6-1. PMID 16426455
- [Background] Pak JG, White SN. Pain prevalence and severity before, during, and after root canal treatment: a systematic review. J Endod. 2011 Apr;37(4):429-38. doi: 10.1016/j.joen.2010.12.016. PMID 21419285
- [Result] Eghbal MJ, Haeri A, Shahravan A, Kazemi A, Moazami F, Mozayeni MA, Saberi E, Samiei M, Vatanpour M, Akbarzade Baghban A, Fazlyab M, Parhizkar A, Ahmadi M, Akbarian Rad N, Bijari S, Bineshmarvasti D, Davoudi P, Dehghan R, Dehghani M, Ebrahimi H, Emami N, Farajian N, Fereidooni R, Ghobadi G, Ghodrati M, Gohari A, Hashemi A, Hosseini M, Karami E, Kheirabadi N, Kozegari S, Labaf Ghasemi H, Majidi A, Malekzadeh P, Mehrabi V, Mohammadi M, Moradi Eslami L, Noghani A, Omatali N, Pourhatami N, Rahbani Nobar B, Rahmani S, Shafaq P, Soofiabadi S, Teimoori S, Vatandoost F, Asgary S. Postendodontic Pain after Pulpotomy or Root Canal Treatment in Mature Teeth with Carious Pulp Exposure: A Multicenter Randomized Controlled Trial. Pain Res Manag. 2020 Jun 30;2020:5853412. doi: 10.1155/2020/5853412. eCollection 2020. PMID 32676136
- [Result] Eren B, Onay EO, Ungor M. Assessment of alternative emergency treatments for symptomatic irreversible pulpitis: a randomized clinical trial. Int Endod J. 2018 Apr;51 Suppl 3:e227-e237. doi: 10.1111/iej.12851. Epub 2017 Oct 16. PMID 28857203
- [Result] Oguntebi BR, DeSchepper EJ, Taylor TS, White CL, Pink FE. Postoperative pain incidence related to the type of emergency treatment of symptomatic pulpitis. Oral Surg Oral Med Oral Pathol. 1992 Apr;73(4):479-83. doi: 10.1016/0030-4220(92)90330-s. PMID 1574311